CLINICAL TRIAL: NCT02282124
Title: Effectiveness of an Advanced Practice Nurse-led Self-management Program on Prevention of Weight Gain, Physical Activity and Medication Adherence in Patients in the First Year After Renal Transplantation
Brief Title: Effectiveness of an APN-led Self-management Program in Patients in the First Year After Renal Transplantation
Acronym: SMP-NEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KEK-ZK-Nr. 2011-0411
Record Dates: First submitted 2014-10-27; First posted 2014-11-04 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Kidney Transplantation; Rental Transplantation
Keywords: weight; self-management; exercise
MeSH Terms: conditions — Body Weight; Motor Activity | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intensity of the intervention follows a defined algorithm during the first eight months after renal transplantation. Behaviours are classified in three groups:
  * Group 1: Patients with optimal behaviour in all three behaviours.
  * Group 2: Patients with slight deviation (defined) from optimal behaviour in one or more behaviours.
  * Group 3: Patients with larger deviation (defined) from optimal behaviour in one or more behaviours.
  All patients (group 1-3) will receive an assessment, education and a monthly reassessment.
  Patients from group 2 und 3 will receive additionally behavioral education and peer involvement. Patients from group 3 will receive additionally a consilium of specialized healthcare professionals such as a nutritionist, physiotherapist, or psychologist.
  Interventions: Behavioral: Self-management program with monthly sessions
- Control (Other)
  Interventions: Behavioral: Usual Care, containing one session

INTERVENTIONS:
Behavioral: Self-management program with monthly sessions — Patients participate in 9 sessions during the first 8th month after transplantaiton
  Arms: Intervention
Behavioral: Usual Care, containing one session — Session takes place within the first three months after transplantation
  Arms: Control

SUMMARY:
The aim of this study is to investigate the effectiveness of the program in patients after renal transplantation using a randomized controlled trial design. Physical, behavioural, and clinical outcomes will be measured at baseline before randomization then 8 and 12 months later.

DETAILED DESCRIPTION:
Renal transplant recipients have to integrate preventive behaviours into their everyday lives. From the literature it is known that patients can only partially adhere to the recommended behaviours. An evidence-based self-management program to support patients in behaviour change was developed with a main focus on prevention of weight gain and increasing physical activity and medication adherence.

The aim of this study is to investigate the effectiveness of the program in patients in the first year after renal transplantation.

The specific aims of this study are:

1. Compare differences in weight gain between subjects in the IG (intervention group) and in the CG (control group).
2. Compare differences in the amount of physical exercise between subjects in the IG group and the CG.
3. Compare differences in self-reported medication adherence between the subjects of the IG group and the CG.

Secondarily, differences in self-reported quality of life, anxiety and depression, and differences in patients' perception of health care provision regarding chronic illness between the subjects of the IG group and the CG will be compared.

Design: Randomised controlled trial, not blinded

Setting and time: The study will take place at the Nephrology Clinic, University Hospital Zürich, from 1 May 2012 through 31 April 2015.

Variables and Measurement: Physical, behavioural, and clinical outcomes will be measured at baseline, before randomization and then 8 and 12 months later. Medication adherence, physical activity, symptoms of depression and anxiety, quality of life and patients' perception of health care provided will be measured with validated questionnaires. Body weight, height, waist to hip ratio and body composition (BCM Fresenius) will be measured at the Nephrology Clinic. Physical activity will be measured with the pedometer StepWatchTM.

Intervention

ELIGIBILITY:
Inclusion Criteria:

* received a kidney or a kidney-pancreas transplant in the University Hospital Zürich

Exclusion Criteria:

* unstable psychiatric disorder
* cognitive impairment
* multi-organ transplantation with lung
* liver or heart
* illiteracy
* not able to speak and understand German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
change from baseline BMI at 8 months | 8th month
  BMI

SECONDARY OUTCOMES:
difference of activity between control and intervention group at month 8 | month 8
  differences in steps measured with pedometer (Stepwatch)
difference of activity between control and intervention group at month 12 | month 12
  differences in steps measured with pedometer (Stepwatch)
change from baseline BMI at 12 months | 12th month
  BMI
difference of self-reported adherence between control and intervention group at month 8 | month 8
difference of self-reported adherence between control and intervention group at month 12 | month 12
change from baseline LTM at 8 months | 8 months
  LTM measured with Body Composition Analysis
change from baseline LTM at 12 months | 12 months
  LTM measured with Body Composition Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spirig, PHD, RN, Principal Investigator — Nursing Director, Head Office of Nursing and Allied Health Professionals
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829